CLINICAL TRIAL: NCT02393547
Title: Lorcaserin for Preventing Weight Gain Among Smokers Receiving Varenicline: A Pilot Study
Brief Title: Lorcaserin for Preventing Weight Gain Among Smokers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ryan T. Hurt, M.D., Ph.D., Associate Professor, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-007240
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Tobacco Use Disorder; Weight Gain
Keywords: obesity
MeSH Terms: conditions — Tobacco Use Disorder; Weight Gain; Obesity | interventions — Varenicline; lorcaserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Varenicline + Lorcaserin (Experimental): Open label all subjects receive both Varenicline and Lorcaserin
  Interventions: Drug: Varenicline; Drug: Lorcaserin

INTERVENTIONS:
Drug: Varenicline — All subjects receive Varenicline
  Other Names: Chantix
Drug: Lorcaserin — All subjects receive Lorcaserin
  Other Names: Belviq

SUMMARY:
This will be an open label clinical trial with all subjects receiving both lorcaserin and varenicline with a primary aim of reducing post cessation weight gain.

DETAILED DESCRIPTION:
This will be an open label clinical trial with all subjects receiving both lorcaserin and varenicline. The investigators will obtain preliminary data on the efficacy of lorcaserin (10 mg twice daily) for 12 weeks in 20 adult weight-concerned cigarette smokers with a BMI of 27 to 40 simultaneously receiving 12 weeks of open-label varenicline and a behavioral intervention to assist with stopping smoking. Secondary aims will be weight, waist circumference, and smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years and ≤65 years of age;
2. smoked ≥10 cigarettes/day for the past 6 months;
3. BMI of 27-40 kg/m2;
4. resides within the Olmsted County area;
5. motivated to stop smoking;
6. weight concerned as shown with the Weight Concern Scale;
7. able to participate fully in all aspects of the study;
8. understood and signed the study informed consent.

Exclusion Criteria:

1. current nonspecific suicidal thoughts or a lifetime history of a suicidal attempt (defined by the Columbia-Suicide Severity Rating Scale [C-SSRS] as a "potentially self-injurious act committed with at least some wish to die, as a result of act.");
2. current moderate or severe depression as assessed by a score of ≥16 on the Center for Epidemiologic Studies-Depression (CES-D);
3. a lifetime history of bipolar disorder or schizophrenia;
4. use of anti-psychotic medication within the past 30 days;
5. use of weight-loss medications within the past 30 days or current participation in a program specifically designed to help with weight loss;
6. weight fluctuations of 20 pounds or more in the past 6 months (self-report);
7. use of any treatments for tobacco dependence within the past 30 days;
8. use of an investigational drug within the past 30 days;
9. recent history (past 3 months) of abuse of or dependence on a substance other than tobacco;
10. current use of benzodiazepines, narcotics, anti-epileptics, or other medications known to interact with lorcaserin (see human subjects section);
11. current use of triptans, monoamine oxidase inhibitors, selective serotonin reuptake inhibitors (SSRIs), selective serotonin-norepinephrine reuptake inhibitors (SNRIs), dextromethorphan, tricyclic antidepressants (TCAs), bupropion, lithium, tramadol, tryptophan, and St. John's Wort, or any other medication known to involve the serotonergic neurotransmitter system (see human subjects section);
12. uncontrolled hypertension (systolic >160 mm Hg and/or diastolic >100 mm Hg) documented on 2 separate occasions;
13. clinically significant acute or chronic progressive or unstable neurologic, hepatic, renal, cardiovascular, respiratory, or metabolic disease;
14. current use of medications known to interact with varenicline or lorcaserin;
15. another household member or relative participating in the study;
16. Known Diabetes;
17. a known allergy to varenicline or lorcaserin;
18. have taken antibiotics within the past 3 months.
19. Women who are pregnant or lactating, or who are of childbearing potential and are likely to become pregnant during the medication phase but are not willing to use a reliable form of contraception, will also be excluded. Reliable forms of contraception include oral contraception, diaphragm or condom (with spermicide), injections, intrauterine device, surgical sterilization, and abstinence.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Hurt, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Hurt RT, Croghan IT, Schroeder DR, Hays JT, Choi DS, Ebbert JO. Combination Varenicline and Lorcaserin for Tobacco Dependence Treatment and Weight Gain Prevention in Overweight and Obese Smokers: A Pilot Study. Nicotine Tob Res. 2017 Aug 1;19(8):994-998. doi: 10.1093/ntr/ntw304. PMID 27852796

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the community surrounding Mayo Clinic (Rochester, MN) between September 2013 and July 2014. Overweight or obese daily smokers who were interested in stopping cigarette use were recruited through the news media and local advertisements in Rochester, MN.
Pre-assignment Details: The current study included an initial telephone screen.After the initial screen, eligible subjects were invited to come for potential enrollment. Visits prior accrual (drug dispensing) included an information meeting (screening, physician physical exam, and informed consent) and baseline visit (screening, baseline measures and drug dispensing).
Period: Overall Study
Arm/Group | Varenicline + Lorcaserin
Started | 20
Completed | 14
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Varenicline + Lorcaserin
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 90.3 (26.2)
Body Mass Index [Mean (Standard Deviation); unit: units on a scale -- kg/m^2] | 30.4 (4.5)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 102.1 (16.0)

OUTCOME MEASURES:

1. Primary Outcome: Post Cessation Weight Change
Description: change in weight from baseline to week 12
Time Frame: 12 weeks
Population: subjects (n=10) who met criteria for prolonged smoking abstinence at week 12
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Varenicline + Lorcaserin
Number analyzed (Participants) | 10
kg | 1.1 (3.9)

2. Secondary Outcome: Waist Circumference
Description: Change in waist circumference from baseline to week 12
Time Frame: 12 Weeks
Population: subjects (n=10) who met criteria for prolonged smoking abstinence at week 12
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Varenicline + Lorcaserin
Number analyzed (Participants) | 10
cm | 0.2 (6.0)

3. Secondary Outcome: Smoking Abstinence Rates
Description: prolonged smoking abstinence at week 12
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline + Lorcaserin
Number analyzed (Participants) | 20
Participants | 10

4. Secondary Outcome: BMI
Description: Change in BMI from baseline to week 12
Time Frame: 12 weeks
Population: subjects (N=10) who met criteria for prolonged smoking abstinence at week 12
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Varenicline + Lorcaserin
Number analyzed (Participants) | 10
kg/m^2 | 0.3 (1.3)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Varenicline + Lorcaserin
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline + Lorcaserin (N=20)
Suicidal Ideation (Psychiatric disorders) | 1 (1) — One serious AE of suicidal ideation was triggered by escalation of marital problems at home and adjudicated not related to the medications.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline + Lorcaserin (N=20)
sleep disturbance (General disorders) | 4 (5) — vivid dreams, sleep disturbance, insomnia
constipation (Gastrointestinal disorders) | 2 (3)
heart burn (Gastrointestinal disorders) | 1 (1)
nausea (General disorders) | 3 (3)
headaches (Nervous system disorders) | 1 (1)
dry mouth (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes